CLINICAL TRIAL: NCT03744806
Title: Blood-aqueous Barrier Integrity in Eyes Undergoing Intravitreal Bevacizumab Therapy to Treat Neovascular Age-related Macular Degeneration
Brief Title: Blood-aqueous Barrier Integrity in Eyes Undergoing Intravitreal Bevacizumab Therapy to Treat Neovascular AMD
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Sponsor
Other Study IDs: KE-0254/208/2013
Record Dates: First submitted 2018-03-22; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Exudative Age-related Macular Degeneration
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- treated with intravitreal bevacizumab.
  Interventions: Drug: Bevacizumab Injection
- control group

INTERVENTIONS:
Drug: Bevacizumab Injection
  Groups: treated with intravitreal bevacizumab.

SUMMARY:
The aim of this study is to evaluate the effect of repeated intravitreal bevacizumab injections on blood-aqueous barrier permeability in eyes with neovascular age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* active AMD-associated choroidal neovascularization (CNV) confirmed with fluorescein angiography (FA) and optical coherence tomography (OCT)

Exclusion Criteria:

* history of uveitis, vitreous hemorrhage, neovascular glaucoma, corneal opacities, recent ocular surgery (within 3 months), or prior anti- vascular endothelial growth factor (VEGF) injections

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Anterior chamber (AC) inflammation evaluated with laser flare photometry. | 4 months
  All patients were examined before and 1 day and 1 month after each intravitreal bevacizumab injection. Subjects were followed for a period of 4 months in both the study and control groups. The final flare photometry value was automatically calculated by averaging 5 individual measurements. A total of 7 measurements were obtained, but the highest and lowest measurement values were excluded by the flare meter. All statistical analyses were performed using STATISTICA 12 statistical software.